CLINICAL TRIAL: NCT05434416
Title: The Efficacy of a Mobile Application in Reducing Craving and Lapse Risk in Alcohol and Stimulants Problematic Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PredictWatch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/001A
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Addiction; Addiction, Alcohol; Addiction, Substance
Keywords: stimulants; alcohol; mobile app; mHealth
MeSH Terms: conditions — Behavior, Addictive; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- No Interventions (No Intervention): Given access to all interventions at the end of the 5 weeks of the trial.
- Short-term interventions (Experimental): Participants have access only to short-term interventions. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Short-term and long-term interventions (Experimental): Short-term and long-term interventions Participants have access to short-term and all long-term interventions.
  Interventions: Other: mobile app
- Long-term intervention: Meditations (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Meditations. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Mindfulness (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Mindfulness. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: My beliefs (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: My beliefs. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Success Diary (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Success Diary. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Gratitude Journal (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Gratitude Journal. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Planner (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Planner. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Journey to Sobriety (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Journey to Sobriety. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Mood Journal (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Mood Journal. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Dream Diary (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Dream Diary. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app
- Long-term intervention: Thinking traps (Experimental): Participants have access to short-term interventions. Participants have access to one long-term intervention: Thinking traps. Given access to all interventions at the end of the 5 weeks of the trial.
  Interventions: Other: mobile app

INTERVENTIONS:
Other: mobile app — mobile app self-guided psychological interventions
  Arms: Long-term intervention: Dream Diary; Long-term intervention: Gratitude Journal; Long-term intervention: Journey to Sobriety; Long-term intervention: Meditations; Long-term intervention: Mindfulness; Long-term intervention: Mood Journal; Long-term intervention: My beliefs; Long-term intervention: Planner; Long-term intervention: Success Diary; Long-term intervention: Thinking traps; Short-term and long-term interventions; Short-term interventions

SUMMARY:
The aim of the study is to evaluate the effectiveness of long-term and short-term app-based self-guided psychological interventions to reduce craving and lapse risk in users with substance use disorder or problematic substance use (alcohol and stimulants). Participants are randomly assigned to thirteen different groups to compare the effectiveness of particular long-term interventions. A questionnaire battery assessment is administered (1) at baseline in the first week following onboarding in; (2) after 5 weeks; (3) after six months. In addition, longitudinal data on several variables related to craving and lapse risk are collected daily using ecological momentary assessment.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of long-term and short-term app-based self-guided psychological interventions to reduce craving and lapse risk in users with substance use disorder or problematic substance use (alcohol and stimulants).

Two main self-guided intervention modules are available. Short-term self-guided intervention module include mainly audio-guided sessions on gratitude, thoughts management, auto-empathy, and relaxation. Moreover, there based on breath relaxation exercises, craving management, and motivation to change Long-term self-guided intervention module include CBT-based interventions, meditations, mindfulness, and journaling.

Participants are recruited via newsletters, local and nation-wide advertisements, as well as through social media. The study is conducted via a mobile application "Nałogometr", freely available to participants. We recruit people from the general population residing in Poland.

To compare the effectiveness of mobile app-based self-guided psychological interventions, participants are randomly assigned to thirteen different groups.

Experimental conditions are balanced based on multiple variables provided during onboarding: (1) main addiction type; (2) participation in addiction-related therapy; (3) gender; (4) age; (5) addiction severity; (6) abstinence duration.

In groups 1-10, participants have access to short-term interventions and one of the long-term interventions. Participants assigned to group 11 have access to short-term and all long-term interventions. Participants in group 12 have access only to short-term interventions. Finally, participants assigned to group 13 serve as the control group and only have access to the weekly ecological momentary assessment reports. However, the control group will be granted access to all intervention materials after five weeks following study enrollment. Participants in group 1-12 will be able to access the intervention materials 5 days after enrollment and will receive weekly ecological momentary assessment reports.

Questionnaire battery assessments will take place: (1) at baseline in the first week following onboarding in; (2) after 5 weeks; (3) after six months. In addition, longitudinal data on several variables related to craving and lapse risk will be collected daily using ecological momentary assessment.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age
* speak Polish fluently
* use either an Android or iOS smartphone

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Lapses rate according to EMA self-report | 5 weeks
  collected daily via the participant's smartphone; an item asking whether or not the lapse occurred since the last survey (yes / no). The score will be tracked for changes over time.
Craving level according to EMA self-report | 5 weeks
  collected daily via the participant's smartphone; an item asking how strong is one's urge to use [substance] at the moment on a scale of 0 to 6 (none - incalculable ). The score will be tracked for changes over time.

SECONDARY OUTCOMES:
Score of Alcohol Use Disorders Identification Test (AUDIT) | 1 week, 5 weeks, 6 months
  Problematic alcohol use will be masured with an Alcohol Use Disorders Identification Test (AUDIT) (WHO, 2001), a 10-item one-dimensional tool. Participant's answer the questions in terms of standard drinks. AUDIT assesses the amount and frequency of alcohol intake (items 1-3), alcohol dependence (questions 4-6), and problems related to alcohol consumption (items 7-10). Questions 1 to 8 are scored on a 5-point scale ranging from 0 to 4, and questions 9 and 10 are scored as 0, 2, or 4. Total scores range from 0 to 40, and the cut-off point to identify hazardous alcohol intake is 8, a score between 16 and 19 indicates harmful alcohol use, and scores above 20 points indicate possible alcohol use disorder.
Score of Severity of Dependence Scale (SDS) | 1 week, 5 weeks, 6 months
  The Severity of Dependence Scale (SDS) (Gossop, et al., 1995) will be used to provide a self-reported measure of psychological aspects of stimulants and alcohol dependence. A five-items, one-dimensional tool has uniform scale for questions 1 - 4 from 0 ('never or almost never') to 3 ('always'). Question 5 has the same scale with different signature where 0 means 'not difficult at all' and 3 means 'impossible'. Score ranging from 0 to 15, where cut-off score depends on user's drug type - a cut-off of =< 3 has been used for indexing alcohol dependence (Lawrinson et al., 2007) and =< 5 for indexing amphetamine dependence (Topp & Mattick, 1997).
Score of Satisfaction With Life Scale (SWLS) | 1 week, 5 weeks, 6 months
  Participants' satisfaction with their life will be assessed with The Satisfaction With Life Scale (SWLS) (Diener et al., 1985), Polish version from Jankowski (2015). SWLS is a short self-report instrument on which participants indicate their agreement to five statements about life satisfaction on a seven-point Likert scale. A maximum score of 35 can be reached, indicating a high level of life satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- PredictWatch, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://badanienalogow.pl/